CLINICAL TRIAL: NCT04409418
Title: Blood Sampling and Extended Dwell Catheters: A Randomized Trial of Blood Sampling Functionality Based on Site Selection
Brief Title: Blood Sampling Functionality of Extended Dwell Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Amit Bahl, Director Emergency Medicine Ultrasound, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-053
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: IV Catheter-Related Infection or Complication; Vascular Access Complication; Peripheral Venous Access
Keywords: intravenous access; vascular access; IV survival

STUDY DESIGN:
Intervention Model Description: Prospective, single-site, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Group (Experimental): If the patient is randomized to the experimental group (lower arm), the research staff will direct the insert to place the catheter into the forearm at least 10 cm away from the antecubital fossa.
  Interventions: Device: Extended dwell catheters
- Control Group (Active Comparator): Control group (upper arm). If the patient is in the control group the research staff will direct the inserter to place the catheter into the upper arm vein at least 2 cm above the antecubital fossa.
  Interventions: Device: Extended dwell catheters

INTERVENTIONS:
Device: Extended dwell catheters — EDCs are generally placed using ultrasound for guidance and are commonly placed in any of 3 veins in the arm. They can be inserted above or below the antecubital fossa (the bend of your elbow). These catheters can be left for up to 30 days and don't fail as quickly when compared to peripheral IVs.

SUMMARY:
The purpose of this study is to compare upper arm versus forearm Extended Dwell Catheter (EDC) placement for blood sampling functionality. EDC is an alternative to peripheral Intravenous (IVs) especially during prolonged hospital stays. EDCs are generally placed using ultrasound for guidance and are commonly placed in any of 3 veins in the arm. They can be inserted above or below the antecubital fossa (the bend of the elbow). These catheters can be left for up to 30 days and don't fail as quickly when compared to peripheral IVs.

DETAILED DESCRIPTION:
Many patients will require ongoing blood draws for laboratory testing while in the hospital and hospitals generally avoid using peripheral IVs for laboratory testing as it is associated with an increase in complications such as irritation and infiltration (where the IV medication or fluid will leak out of the vein and into the surrounding tissue). Therefore, patients are often required to have multiple needlesticks throughout their hospital stay which can lead to patient dissatisfaction and anxiety.

Extended dwell catheters (EDC) offer an alternative to peripheral IVs especially during prolonged hospital stays. EDCs are generally placed using ultrasound for guidance and are commonly placed in any of 3 veins in the arm. They can be inserted above or below the antecubital fossa (the bend of the elbow). These catheters can be left for up to 30 days and don't fail as quickly when compared to peripheral IVs. While there is not a lot of evidence about how well these catheters will allow blood to be drawn, an EDC can be used to obtain blood for routine blood draws and potentially eliminate the need for additional needle sticks.

Eligible patients in this study will be randomized to two groups based on placement site: experimental group (forearm) or the control group (upper arm). If the patient is in the control group the research staff will direct the inserter to place the catheter into the upper arm vein at least 2 cm above the antecubital fossa. If the patient is randomized to the experimental group (lower arm), the research staff will direct the insert to place the catheter into the forearm at least 10 cm away from the antecubital fossa. The research team will capture images on the ultrasound machine that is used for initial assessment of sites per routine care. If the vein is appropriate for cannulation based on these assessments, the Advance Practice Provider (APP) will insert the catheter. If the APP on the Vascular Access Team (VAT) has no adequate target visualized in the randomly selected site, the inserter may evaluate another site that is more suitable for cannulation. Functionality will be confirmed by ability to aspirate by drawing back into a syringe and then the catheter flushed with 5cc of normal saline without resistance. The site of insertion will be recorded and pertinent information will be collected similar to other catheter placements. Securement of the placed IV will be standardized between groups. Daily assessment of functionality (patency of the catheter) will be performed by the research team for the life of the catheter while hospitalized (up to 30 days).

ELIGIBILITY:
Inpatient Inclusion Criteria:

1. Consult to VAT for vascular access device placement
2. Patient requires peripheral access
3. Adults >18 years of age

ED Patient Inclusion Criteria

1. Age > 18 years old
2. Difficult vascular access defined as: patient has no visible veins (>2mm) or palpable veins
3. Anticipated hospital admission

All patients meeting inclusion criteria will be pre-scanned prior to formal enrollment to identify diameter of target veins and calculate a catheter to vein ratio at the potential insertion site. Patients must meet this criteria in both upper arm and forearm locations prior to enrollment and randomization.

Exclusion Criteria:

Patients will be excluded if:

1. Multiple lumens required
2. Functional vascular access device exists proximal to the targeted area of insertion. This does not include superficial non-ultrasound guided peripheral IVs.
3. Upper extremity cannot be accessed due to a coexisting medical condition
4. Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 100 were consented. Prior to randomization, 9 patients were excluded for inadequate vessel size, 2 patients withdrew from the study, 1 patient investigator removed due to other IV access.
  20 patients originally assigned to the forearm group crossed over to the upper arm group because there was no suitable target vessel, leaving 24 in the forearm group and 64 in the upper arm group.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 24 | 64
Completed | 24 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 24 | 64 | 88
Age, Customized [Count of Participants; unit: Participants]
  <=25 years | 2 | 1 | 3
  26-50 years | 4 | 14 | 18
  51-75 years | 13 | 34 | 47
  >75 years | 5 | 15 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 39 | 50
  Male | 13 | 25 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 64 | 88

OUTCOME MEASURES:

1. Primary Outcome: Blood Sampling Functionality
Description: Blood sampling ability will be evaluated by daily blood draws prior to patient discharge. The measured outcome is number of hours until failure to aspirate blood identified during follow-up assessment during hospitalization.
Time Frame: During hospitalization, up to 30 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 24 | 64
hours | 70.19 (61.41) | 112.9 (141.47)

2. Secondary Outcome: Catheter Dwell Time/Survival
Description: Functionality of catheter for intravenous therapy prior to patient discharge. The measured outcome is number of hours until failure of functionality identified as inability to infuse without resistance during follow-up assessment during hospitalization.
Time Frame: During hospitalization, up to 30 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 24 | 64
hours | 74.27 (59.9) | 115.52 (140.42)

3. Secondary Outcome: Thrombosis
Description: The number of participants with symptomatic catheter-related upper extremity venous thrombosis (CR-UEVT) inclusive of superficial thrombophlebitis (SVT) and deep venous thrombosis (DVT) confirmed by upper extremity venous duplex evaluation.
Time Frame: During hospitalization, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 24 | 64
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: During hospital admission (beginning at enrollment) through 30 days post discharge, an average of 40 days
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/64
Other Adverse Events (participants affected / at risk) | 6/24 | 24/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=24) | Control Group (N=64)
Catheter occlusion (Product Issues) | 3 (3) | 13 (13)
Infiltration (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Catheter dislodgement (Product Issues) | 1 (1) | 3 (3)
Catheter leakage (Product Issues) | 1 (1) | 2 (2)
Superficial vein thrombosis (Vascular disorders) | 2 (2) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT04409418/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT04409418/ICF_001.pdf